CLINICAL TRIAL: NCT05894161
Title: Efficacy of Designed Exercise Program on Pain and Quality of Sleeping in Patient With Sickle Cell Disease Anemia.
Acronym: SCDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Eyad Alshurafa, ealshurafa, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-UGS-2022-03-186
Record Dates: First submitted 2023-05-22; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
Keywords: sleep disturbance; Fatigue; Stress; Quality of life
MeSH Terms: conditions — Anemia, Sickle Cell; Parasomnias; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: To prevent human bias regarding to participants and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-I (Experimental): Group-1: Twenty-five adult patients with SCD will receive a designed exercise program of physical therapy for relief pain and improve sleep quality (experimental group). The designed exercise program will be distributed on everyone. The recommendations will be to train from 30 to 45 minutes, 3 days per week for 6 weeks in addition to walking 30 minutes on the ground surface daily.
  Interventions: Other: Exercise training program
- Group-II (No Intervention): Group-2: Twenty-five adult patients with SCD will participate as a control group they will not receive exercise program.

INTERVENTIONS:
Other: Exercise training program — The designed exercise program will be distributed on everyone. The recommendations will be to train from 30 to 45 minutes, 3 days per week for 6 weeks in addition to walking 30 minutes on the ground surface daily.
  1. Diaphragmatic Breathing Exercises: Diaphragmatic breathing (DBRT) or abdominal deep breathing is an expansion of the abdominal area rather than the thoracic area when breathing.
  2. Progressive Muscle Relaxation (PMR): The physical element includes the tensing and relaxing of all muscle groups over the face, arms, trunk (abdomen & chest) and legs.
  3. A combination of stretching, stabilization and strengthening exercises of the pelvic-lumbar region:
  4. Walking exercise: Walking on the ground surface for 30 minutes every day.
  Arms: Group-I

SUMMARY:
Background: Pain and sleep disturbance are the most common problems experienced by adult patients with sickle cell disease anemia. Aim: the aim of this study is to evaluate the efficacy of designed exercise program on pain, and quality of sleeping in adult patients with sickle cell disease anemia and how the program affects their quality of lives. Subjects and methods: Adults patients with sickle cell diseases aging over 18 years old. Data will be collected in face-to-face interviews. Eligible participants will be equally and randomized into two groups. Group-1: Twenty-five adult patients with SCD will receive a designed exercise program of physical therapy for relief pain and improve sleep quality (experimental group). The designed exercise program will be distributed on everyone. The recommendations will be to train from 30 to 45 minutes, three days per week for 6 weeks in addition to walking daily 30 minutes on the ground surface. Group-2: Twenty-five adult patients with SCD will participate as a control group they will not receive exercise program. Analysis: The collected data will be managed by using t -test and the repeated measures of ANOVA test to compare the significance within groups and between two groups.

DETAILED DESCRIPTION:
Methodology:

Design: Randomized clinical trial (RCT). Subjects' criteria: Fifty adult sickle cell disease patients who are aged more than 18 years with different socio-economic and educational levels. Patients with sickle cell anemia will be distributed into two groups. All personal data will be collected.

Group-1: Twenty-five adult patents with SCD will receive a designed exercise program of physical therapy for relief pain and improve sleeping quality (experimental group). The designed exercise program will be distributed on everyone. The recommendations will be to train from 30 to 45 minutes, three days per week for 6 weeks in addition to walking daily 30 minutes on the ground surface.

Group-2: Twenty-five adult patients with SCD will participate as a control group they will not receive exercise program.

Assessment instruments:

1. Pittsburgh Sleep Quality Index: The (PSQI) is a 19-item instrument created to measure different aspects of sleep quality and sleep disturbance (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). The scale reports quality of sleeping over the past month. The PSQI is divided into 7 subscale scores: subjective sleep quality; sleep latency (time of full sleep); duration; habitual sleep efficiency (proportion between total sleep time and time in bed); sleep disturbances (waking up during the night); use of medication to sleep; and daytime dysfunction (difficulty staying awake during daytime). The overall score ranges between 0 and 21, and a total score of more than 5 indicates poor sleep quality(Al Maqbali et al., 2020).
2. WHOQOL-BREF: The World Health Organization (WHO) identified Quality of Life (QoL) as "an individual's perception of his or her position in life, within the context of the culture and value systems in which they live, and in regard to his or her goals, expectations, standards and concerns" . QoL is consist of multiple aspects, including psychological health, physical well-being, social relationships, and environmental conditions. Although health professionals are trained on attending to these aspects during studies, own QoL might decline during the years in medical schools(Bani-Issa, 2011).
3. Visual Analog Scale: VAS: It is a safe, valid, and reliable measurement instrument used to evaluate pain severity. It was designed by Huskisson to quantify values that could not be measured in numbers. The most important advantage of the test is the lack of a language barrier and simplicity of application. The definition of the parameter to be assessed is written at the two ends of a 10 cm line, and the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks (Kazak and Ozkaraman, 2021, Crichton, 2001).

4 - The Fatigue Scale: The fatigue scale, established by Chalder etal., is choosing to study the incidence of fatigue. The scale contains 11 questions, seven physical and four mental fatigue items. Patients will be asked if they had suffered each symptom in the last two weeks and the scale will be scored using a bimodal response system (0,0,1,1). the fatigue score will be calculated by adding together all the item scores (maximum score 11) and the total of four or more constituted a case of fatigue (Mcllvenny, 1999).

5 - The Perceived Stress Scale: The (PPS) has been designed to measure the degree to which situations in a person's life are perceived as stressful. The PSS assesses the level of perceived stress experienced over the previous month, and has three versions: the PSS-14, PSS-10 and PSS-4 with 14 and 10 and 4 items respectively. The PSS-14 has seven positive and seven negative items. The Arabic version Perceived Stress Scale showed an adequate reliability and validity. Therefore, the Arabic Perceived Stress Scale is considered a suitable instrument to assess perceived stress in Arabic people (Almadi et al., 2012).

Randomization type is blocking randomization. It will be taken by the main researcher using a random number generator by computer program software http://mahmoodsaghaei.tripod.com/Softwares/randalloc.html#Generate.

Ethical approval: It will be obtained from the Institutional Review Board (IRB) at Imam Abdulrahman Bin Faisal University.

Confidentiality: All data of participants will be saved in a personal computer locked with a password. All questionnaires' papers will be kept with the main researcher in a locker.

Patient's rights: All recruited patients will sign a consent form before their participation, and they will be informed that the collected data will be published.

Inclusion criteria: SCD patient, aged < 18 years, have no communication problems, did not regularly perform relaxation exercises, and able to perform the exercises.

Exclusion criteria: Patients with SCD who are aged less than 18, unable to do the exercises and had communication problems.

Procedures of the study:

Fifty adult patients with SCD, will be randomly assigned to either experimental or control group. All patients will receive face-to-face instructions and explanations about the procedure of the study and assessment tools. The training period will take 6 weeks (details pertaining to the program which will be specified below) and the post-test including the same measures of the VAS, PSQI, WHOQOL-BREF, The Fatigue Scale and The PSS at the end of the 6-week program.

Group-I: Every patient will practice on exercise program for 30 to 45 minutes day other day for 6 weeks. All patients in the first group will participate as experimental group who will receive a designed exercise program of physical therapy for relief pain and improve sleep quality. They will be provided with a manual containing the necessary guidelines of the exercises and instructions to train from 30 to 45 minutes in addition to walking 30 minutes daily on the ground surface for 3 days per week for 6 weeks. The pre and post measurements will be done for all patients.

Group-II: All patients of the second group will participate as a control group, they will not participate in the exercise program but the pre and post measurements will be done for all patients.

Interventions:

Group-1: Twenty-five adult patients with SCD will receive a designed exercise program of physical therapy for relief pain and improve sleep quality (experimental group). The designed exercise program will be distributed on everyone. The recommendations will be to train from 30 to 45 minutes, 3 days per week for 6 weeks in addition to walking 30 minutes on the ground surface daily.

1. Diaphragmatic Breathing Exercises: Diaphragmatic breathing (DBRT) or abdominal deep breathing is an expansion of the abdominal area rather than the thoracic area when breathing. Diaphragmatic breathing is a manipulation of breath movement that contributes to a physiological response(Jerath et al., 2006). The benefits of DBRT have been demonstrated by Stromberg et al. (Stromberg et al., 2015) and Aslan et al. (Aslan et al., 2016). They explained that DBRT is an effective non-pharmacological treatment for improving sleep and emotions, resulting in diminished levels of anxiety, depression, and stress. And deep breathing has been shown to cause cardiopulmonary synchronization, resulting in stronger sympathetic inhibition. In contrast, fast or irregular breathing can lead to sympathetic excitation(Liu et al., 2021).
2. Progressive Muscle Relaxation (PMR): The physical element includes the tensing and relaxing of all muscle groups over the face, arms, trunk (abdomen & chest) and legs. In a sequential pattern, with eyes closed. Every patient places a tension in each muscle group purposefully for approximately 10 seconds and then relaxes it for 20 seconds before continuing with the next muscle group. The mental element involves that the individual concentrates on the distinction between the feelings of the tension and relaxation. Every patient with practice learns how to successfully relax in a short period of time. Relaxation must be attempted to reduce pain or pain perception and tension, create a pleasant mental state. The exercise will be performed in an average of 30 minutes. The PMR sessions will be performed in a comfortable armchair(Benson et al., 1974, Örsal et al., 2014).
3. A combination of stretching, stabilization and strengthening exercises of the pelvic-lumbar region: The exercises will be performed 3 times a week, three repetitions for 30 seconds:

   Exercise 1 - Unilateral flexion of the lower limbs over the abdomen:

   Aim: Bilateral stretching of one side of the lower quarters and for the upper quarter of the opposite side (lumbo-pelvic region), time: 30 seconds, repetitions: 3.

   Exercise 2 - Lower limb flexion over the abdomen:

   Aim: Stretching and stabilization of the lumbo-pelvic region, time: 30 seconds, repetitions: 3.

   Exercise 3 - Knee Roll:

   Aim: Strengthens medial rotators (tensor fascia lata muscle, gluteus minimus and gluteus medius and laterals -pyriform, femoral quadrate, internal and external obturators, superior and inferior gemelli) of the hip, time: 30 seconds, repetitions: 3.

   Exercise 4 - Bridge:

   Aims: Improves gluteus strength and strength of the muscles in the posterior thigh; Stretching of the flexor muscles of the hip (ilio-psoas and quadriceps); Improves lumbo-pelvic stability (torso and hips); Improves backbone mobility, time: 30 seconds repetitions: 3.

   Exercise 5 - Hyperextension of the hip moving against gravity:

   Aim: Strengthening of the extensor muscles of the hip (muscles of the gluteal regions and of the posterior thigh), time: 30 seconds, repetitions: 3 (Zanoni et al., 2021).
4. Walking exercise: Walking on the ground surface for 30 minutes every day. Group-2: Twenty-five adult patients with SCD will participate as a control group they will not receive exercise program.

Statistical analysis: the T-test and repeated measure analysis of ANOVA will be used to compare mean values within and between two groups. Results will be significant at P-value < 0.05 and confidence interval at 0.95 %.

ELIGIBILITY:
Inclusion Criteria:

1. SCD patient
2. Their age from18 -55 years
3. have no communication problems
4. They able to perform the exercises

Exclusion Criteria:

1. Their age less than 18
2. They unable to do the exercises.
3. They had communication problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 10 minutes
  The (PSQI) is a 19-item instrument created to measure different aspects of sleep quality and sleep disturbance (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). The scale reports quality of sleeping over the past month. The PSQI is divided into 7 subscale scores: subjective sleep quality; sleep latency (time of full sleep); duration; habitual sleep efficiency (proportion between total sleep time and time in bed); sleep disturbances (waking up during the night); use of medication to sleep; and daytime dysfunction (difficulty staying awake during daytime). The overall score ranges between 0 and 21, and a total score of more than 5 indicates poor sleep quality(Al Maqbali et al., 2020).
Visual Analog Scale: | 5 minutes
  VAS: It is a safe, valid, and reliable measurement instrument used to evaluate pain severity. It was designed by Huskisson to quantify values that could not be measured in numbers. The most important advantage of the test is the lack of a language barrier and simplicity of application. The definition of the parameter to be assessed is written at the two ends of a 10 cm line, and the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks (Kazak and Ozkaraman, 2021, Crichton, 2001).

SECONDARY OUTCOMES:
WHOQOL-BREF: | 5 minutes
  The World Health Organization (WHO) identified Quality of Life (QoL) as "an individual's perception of his or her position in life, within the context of the culture and value systems in which they live, and in regard to his or her goals, expectations, standards and concerns" . QoL is consist of multiple aspects, including psychological health, physical well-being, social relationships, and environmental conditions. Although health professionals are trained on attending to these aspects during studies, own QoL might decline during the years in medical schools(Bani-Issa, 2011).
The Fatigue Scale | 5 minutes
  The fatigue scale, established by Chalder etal., is choosing to study the incidence of fatigue. The scale contains 11 questions, seven physical and four mental fatigue items. Patients will be asked if they had suffered each symptom in the last two weeks and the scale will be scored using a bimodal response system (0,0,1,1). the fatigue score will be calculated by adding together all the item scores (maximum score 11) and the total of four or more constituted a case of fatigue (Mcllvenny, 1999).
The Perceived Stress Scale | 3 minutes
  The (PPS) has been designed to measure the degree to which situations in a person's life are perceived as stressful. The PSS assesses the level of perceived stress experienced over the previous month, and has three versions: the PSS-14, PSS-10 and PSS-4 with 14 and 10 and 4 items respectively. The PSS-14 has seven positive and seven negative items. The Arabic version Perceived Stress Scale showed an adequate reliability and validity. Therefore, the Arabic Perceived Stress Scale is considered a suitable instrument to assess perceived stress in Arabic people (Almadi et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Alsayed Shanb, Phd, Study Director — Associate professor in CAMS in IABF university
Locations (1):
- IAU, Dammam, Estern, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
General data not individualized